CLINICAL TRIAL: NCT01504880
Title: Evaluation of Mitral and Tricuspid Regurgitation: Cardiovascular Magnetic Resonance Imaging Versus Echocardiographic Doppler Color Flow Mapping of the Vena Contracta
Brief Title: Atrioventricular Valve Regurgitation Vena Contracta; Echo Versus MRI
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Benjamin Goot, Assistant Professor, Pediatrics, Cardiology, Medical College of Wisconsin
Other Study IDs: CHW 09/155; GC 960 (Other: Medical College of Wisconsin)
Record Dates: First submitted 2012-01-03; First posted 2012-01-06 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Tricuspid Valve Regurgitation, Non-rheumatic; Mitral Valve Regurgitation
Keywords: Mitral Regurgitation; Tricuspid Regurgitation; Vena Contracta
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this pilot study is to evaluate mitral (left atrioventricular valve) and tricuspid (right atrioventricular valve (AVV)) regurgitation using cardiac magnetic resonance imaging (CMR) as the non-invasive "gold standard" compared to transthoracic echocardiography (TTE) to evaluate measurements of the width of the regurgitation jet (vena contracta (VC)) to demonstrate the utility of the VC as a means to objectively evaluate atrioventricular valve regurgitation. In addition, feasibility and other quantitative and qualitative measures of regurgitation will be compared between CMR and TTE.

* Hypothesis 1: The ability to objectively evaluate atrioventricular valve regurgitation and VC width with TTE and CMR has a high feasibility rate with acceptable intra and inter-observer variability by two independent readers.
* Hypothesis 2: There will be positive correlation between the TTE measurement of the VC width and quantitative assessment of atrioventricular valve regurgitation by TTE and CMR.
* Hypothesis 3: There will be a positive correlation between the quantitative measurements of atrioventricular valve regurgitation by phase contrast velocity encoded CMR with quantitative values as measured by TTE.
* Hypothesis 4: There will be a positive correlation between qualitative assessment of atrioventricular valve regurgitation by CMR compared to TTE.

DETAILED DESCRIPTION:
BACKGROUND, SIGNIFICANCE, AND RATIONALE (including preliminary studies and any results) The integrity of the two atrioventricular valves (AVV)(i.e., the mitral and tricuspid valve) plays an important role in the evaluation and management of patients with congenital and acquired heart disease. Loss of valve integrity (i.e., valve leakage in the reverse direction of normal blood flow), is known as valve regurgitation. Increasing severity of mitral regurgitation has been associated with increased mortality and morbidity. Tricuspid regurgitation can be a progressive problem that results in right atrial and ventricular dilation and possible right heart failure. Similarly, mitral valve regurgitation can result in left atrial and left ventricular enlargement. Treatment options for valvular regurgitation are based upon the degree of regurgitation in both adults and children. Therefore, assessment of the degree of AV valvular regurgitation has important clinical ramifications. AV valve regurgitation can be assessed in several ways, including both invasive and noninvasive modalities. The invasive assessment is performed by cardiac catheterization which enables qualitative and quantitative measurements of AV valve regurgitation and in the past has been considered the "gold standard". Noninvasive assessment is still the preferred method and consists of echocardiography, electrocardiography, chest x-ray, and CMR. TTE can be used qualitatively to describe the amount of AV valve regurgitation by the degree of color flow Doppler reflux into the left atrium during left ventricular contraction. This approach grades the regurgitation as mild, moderate or severe similar to angiographic grading systems, but is relatively subjective and affected by technical factors. TTE can quantitatively evaluate AV valve regurgitation through calculation of regurgitation orifice area, regurgitation volume and regurgitation fraction. These methods have been shown to have a good correlation when used for mitral valves compared to cardiac catheterization and CMR in adults. However, quantitative techniques are time consuming and require multiple measurements and more complex calculations. A simpler technique of objectively characterizing the regurgitation of the AV valves by TTE is measuring the width of the vena contracta (VC). The VC is the narrowest portion of a regurgitant jet which occurs at the level of or just below the valve leaflets and represents the effective regurgitant orifice. In adult studies, this method has shown that increase in VC width of the mitral valve strongly correlates with qualitative angiographic grades and quantitative measurements of regurgitant volume by cardiac catheterization and is a better assessment of regurgitation than measuring the regurgitant jet by TTE. Changes in VC width also had strong correlation with quantitative measurements of regurgitant volume and regurgitant orifice area using TTE. It is our intent to evaluate the feasibility and correlation of measurements of AV valve regurgitation by TTE with focus on the VC in pediatric patients compared to the non-invasive "gold standard" measurements by CMR.

ELIGIBILITY:
Inclusion Criteria:

* Audible AV valve regurgitation on clinical exam, as noted by most recent clinic note.
* Clinically indicated CMR study scheduled and have had an echocardiogram in the last 6 months

Exclusion Criteria:

* Poor quality CMR study
* Unable to complete a CMR
* Have a contraindication to CMR scan (e.g., pregnancy, pacemaker or defibrillator presence, unable to hold still within scanner for imaging)
* Common AV valve
* Corresponding semilunar valve regurgitation which precludes use of stroke volume comparison as a second means of assessing AVV regurgitation by CMR
* Intracardiac shunts which precludes use of stroke volume comparison as a second means of assessing AVV regurgitation by CMR.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for clinically indicated MRI and have had an echocardiogram in the last 6 months with AV Valve (AVV) Insufficiency.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-06; Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Vena Contracta Value | At time of Echo and MRI
  Comparison of the echocardiographic measured vena contracta with quantitative value of mitral or tricuspid regurgitation as measured by MRI.

SECONDARY OUTCOMES:
Mitral and Tricuspid Regurgitation Fraction | At time of Echo and MRI
  Quantitative echo measurements of mitral or tricuspid valve regurgitation fraction will be correlated to MRI derived regurgitation fraction of the mitral or tricuspid valves.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Goot, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes